CLINICAL TRIAL: NCT03091647
Title: Acupressure Intervention to Improve Fatigue and Physical Functioning of Chinese Immigrant Breast Cancer Survivors
Brief Title: Acupressure for Cancer-Related Fatigue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Judy Wang, Associate Professor, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-0435
Record Dates: First submitted 2017-03-17; First posted 2017-03-27 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
Keywords: Chinese women; Cancer-related fatigue; Acupressure
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupressure intervention (Experimental): Practice acupressure at home and complete daily logs
  Interventions: Behavioral: acupressure intervention
- usual care (Placebo Comparator): Receive usual care and complete daily logs
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: acupressure intervention — Women in the acupressure intervention group will learn how to press three chief energy acupoints on each side of the body through an 11-minute Chinese-language video and press three acupoints (1 minute per acupoint) on both sides of the body every day for a total of 6 minutes per day for an 8-week intervention period and record their practice on daily logs. Women will be asked to return the logs every week by email or self-addressed envelopes.
  Arms: acupressure intervention
Behavioral: usual care — Women in the usual care group will receive primary and oncology care from their doctors as usual, and complete daily logs recording their fatigue and daily functioning levels. They also need to return the logs every week by email or self-addressed envelopes.
  Arms: usual care

SUMMARY:
This study develops and pilot tests the efficacy of a home-based, self-administered acupressure intervention in improving cancer-related fatigue (proximal outcome), and physical functioning and other quality of life outcomes (distal outcomes) of Chinese immigrant breast cancer survivors (versus usual care control group).

DETAILED DESCRIPTION:
We will enroll 124 foreign-born, Chinese-speaking women from Southern California and Maryland areas with moderate to severe levels of fatigue, diagnosed with stage 0-IV breast cancer, aged 21-74, and 1-5 years post-primary treatment. Using an adaptive treatment strategy design, participants will be randomized to either the acupressure intervention or control groups. The acupressure group will learn how to press three chief energy acupoints on each side of the body through de novo 11-minute Chinese-language video and practice acupressure every day (one minute per acupoint; a total of 6 minutes per day) for an 8-week intervention period. Participants will be telephone interviewed twice: at baseline and 8-weeks post-intervention follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 1) be between ages 21 to 74
* 2) be first-generation immigrants
* 3) speak Chinese (Mandarin and/or Cantonese)
* 4) be diagnosed with breast cancer at stage 0, I, II III or IV
* 5) have completed primary treatments (including surgery, radiation, and chemotherapy) 1-5 years prior to recruitment
* 6) have not had recurrence
* 7) have moderate to severe levels of fatigue.

Exclusion Criteria:

* have hypothyroidism and anemia
* being using acupuncture

Ages: 21 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Cancer-related fatigue (proximal outcome) | 8 weeks post-intervention
  The primary outcome will be measured by 6-item PROMIS (Patient-Reported Outcomes Measurement Information System) (e.g., felt tired, exhausted, limited at work).

SECONDARY OUTCOMES:
Physical functioning (distal outcomes) | 8 weeks post-intervention
  The secondary outcomes will be measure by 8-item PROMIS (e.g., ability in carrying grocery, kneeling, climbing stairs).
Sleep disturbance | 8 weeks post-intervention
  The secondary outcomes will be measure by 6-item PROMIS (e.g., sleep not steady, unsatisfied, hard to fall asleep).
Anxiety | 8 weeks post-intervention
  The secondary outcomes will be measure by 7-item PROMIS (e.g., felt anxious, nervous, fearful, tense).
Depression | 8 weeks post-intervention
  The secondary outcomes will be measure by 8-item PROMIS (e.g., felt helpless, depressed, unhappy, hopeless).
Pain interference | 8 weeks post-intervention
  The secondary outcomes will be measure by 6-item PROMIS (e.g., affecting ability to focus, interact with others, run errands).

CONTACTS AND LOCATIONS:
Overall Officials: Judy Wang, Ph.D., Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided